CLINICAL TRIAL: NCT02786095
Title: Comparison Study of Drugs for Symptom Control and Complication Prevention of Atrial Fibrillation (AF) (Code-AF Trial)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2016-0105
Record Dates: First submitted 2016-05-25; First posted 2016-05-30 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; anti arrhythmic drug; NOAC; warfarin; coumadin
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Code-AF registry

SUMMARY:
This study is prospective Cohort study which was performed in multicenter (General Hospital) in Korea. Inclusion criteria is all patients with atrial fibrillation who visit hospital. The purpose is to analyze complication, composite outcome (all cause mortality, hospitalization, the incidence of stroke, heart failure and cardiovascular event (MACE)) according to the 1) the use of anti-arrhythmic drugs (AADs), 2) use of medication for rate control (beta blocker, calcium channel blocker and digoxin) and 3) use of anticoagulation agents (warfarin, coumadin, an NOAC)

ELIGIBILITY:
Inclusion Criteria:

* patients with atrial fibrillation
* patients with age more than 19
* patients who agree with study inclusion

Exclusion Criteria:

* patients who do not agree with study inclusion
* patients with age less than 19
* Pregnancy, Breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | 3 years
number of hospitalization by heart failure | 3 years
number of recurrent stroke | 3 years
number of cardiovascular events | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Yonsei University Health System, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park H, Yu HT, Kim TH, Park J, Park JK, Kang KW, Shim J, Kim JB, Kim J, Choi EK, Park HW, Lee YS, Joung B. Oral Anticoagulation Therapy in Atrial Fibrillation Patients with Advanced Chronic Kidney Disease: CODE-AF Registry. Yonsei Med J. 2023 Jan;64(1):18-24. doi: 10.3349/ymj.2022.0455. PMID 36579375
- [Derived] Kim JY, Park HS, Park HW, Choi EK, Park JK, Kim JB, Kang KW, Shim J, Joung B, Park KM. Clinical Outcomes of Rhythm Control Strategies for Asymptomatic Atrial Fibrillation According to the Quality-of-Life Score: The CODE-AF (Comparison Study of Drugs for Symptom Control and Complication Prevention of Atrial Fibrillation) Registry. J Am Heart Assoc. 2022 Sep 20;11(18):e025956. doi: 10.1161/JAHA.122.025956. Epub 2022 Sep 8. PMID 36073646
- [Derived] Kim M, Kim J, Kim JB, Park J, Park JK, Kang KW, Shim J, Choi EK, Lee YS, Park HW, Joung B. Association of Gender With Clinical Outcomes in a Contemporary Cohort of Patients With Atrial Fibrillation Receiving Oral Anticoagulants. Korean Circ J. 2022 Aug;52(8):593-603. doi: 10.4070/kcj.2021.0399. Epub 2022 Apr 26. PMID 35656931
- [Derived] Lee KB, Kim TH, Park J, Park JK, Kang KW, Kim J, Park HW, Choi EK, Kim JB, Lee YS, Shim J, Joung B. Stroke and Systemic Thromboembolism according to CHA2DS2-VASc Score in Contemporary Korean Patients with Atrial Fibrillation. Yonsei Med J. 2022 Apr;63(4):317-324. doi: 10.3349/ymj.2022.63.4.317. PMID 35352882